CLINICAL TRIAL: NCT06406231
Title: Magnetic Field Therapy Versus Transcutaneous Electrical Nerve-stimulation in Knee Osteoarthritis: a Head-to-head Trial
Brief Title: Magnetic Field Therapy Versus Transcutaneous Electrical Nerve-stimulation in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, RAZGALLAH Emna, medical resident, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35/2023/CLPP
Record Dates: First submitted 2024-05-05; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Patients treated with transcutaneous electrical nerve stimulation (TENS) (Active Comparator)
  Interventions: Device: comparing efficacy of TENS and PEMF in knee osteoarthritis
- Group 2: Patients treated with magnetotherapy (PEMF) (Active Comparator)
  Interventions: Device: comparing efficacy of TENS and PEMF in knee osteoarthritis

INTERVENTIONS:
Device: comparing efficacy of TENS and PEMF in knee osteoarthritis — Sessions will be conducted by a physiotherapist from the center, trained in the technique.Three sessions per week for three weeks. We used an Automatic Program (approximately 20 minutes).
  For each group, the physical therapy was given as below:
  G2: Patients treated with magnetotherapy:
  -Device used: a prototype of a Health magnetic therapy (H.M.T) generator developed by a group of engineering researchers at the University of Tunis El Manar, employing low-frequency electromagnetic waves. The chosen program is "Analgesia". An applicator containing magnets will be placed on the affected knees. The patient will sit on a chair bending knees.
  G1 : Patients treated with TENS
  -Device used: TENS from ECO2 from Schwa Medico, 2016, France. We chose the "Gate control" program (high frequency). The patient will sit with bent knees on a chair and adhesive patches will be placed on the affected knee. The intensity will be adapted to the patient's tolerance in both groups.

SUMMARY:
The effectiveness of PEMF in improving physical function among Osteoarthritic (OA) patients remains a topic of debate, leading to the American College of Rheumatology not yet endorsing its use in OA treatment. Therefore, it's essential to investigate PEMF therapy's efficacy in alleviating joint pain, stiffness, and enhancing physical function in knee OA patients Our study objectives were to evaluate the effectiveness and safety of PEMF therapy and to compare its efficacy with TENS in knee OA management.

ELIGIBILITY:
Inclusion Criteria:

* We included patients who had knee pain due to knee OA diagnosed according to the American College of Rheumatology including:
* Knee pain AND presence of at least three of the following 6 criteria:

  * Age > 50 years
  * Morning stiffness < 30 minutes
  * Crepitus during movement
  * Periarticular bone pain
  * Periarticular bone hypertrophy
  * Absence of increased local warmth.

Exclusion Criteria:

* For both groups, we did not include:

  * Patients with a pacemaker, implantable defibrillator, cochlear implant, or any metal implant contraindicating MRI (knee prosthesis, hip prosthesis, etc.).
  * Pregnant women
  * Patients with an active infection
  * Profound hypoesthesia or thermoalgic sensitivity disorder
  * Poorly vascularized areas: arteritis, phlebitis, ischemia
  * Patients on anti-vitamin K treatment or with a coagulation disorder. Patients with long-term corticosteroid therapy or having a total knee replacement, those who have received therapies for knee osteoarthritis including intra-articular corticosteroid injection or viscosupplementation in the last 4 months, and Patients with knee pain of non-osteoarthritic origin were also not included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
response to physical therapy | one week before the beginning and 3 weeks after the finishing of the rehabilitation program
  a 20 percent decrease in the total score of WOMAC pain

SECONDARY OUTCOMES:
reduction of pain | one week before the beginning and 3 weeks after the finishing of the rehabilitation program
  Reduction in visual analog scale (VAS) pain scores at rest and during activity.
Consumption of paracetamol | one week before the beginning and 3 weeks after the finishing of the rehabilitation program
assessing safety | one week before the beginning and 3 weeks after the finishing of the rehabilitation program
  occurrence of adverse effects requiring temporary or permanent discontinuation of the technique.
assessing patients satisfaction | one week before the beginning and 3 weeks after the finishing of the rehabilitation program
  Satisfaction VAS
stiffness and function improvement | one week before the beginning and 3 weeks after the finishing of the rehabilitation program
  • Improvement in all three domains of WOMAC and overall WOMAC score: Stiffness (2 questions) and function (17 questions) WOMAC subscales

CONTACTS AND LOCATIONS:
Locations (1):
- Military Hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided